CLINICAL TRIAL: NCT02952170
Title: The Impact of Weight Loss Surgery in Adolescents on Fatty Liver Disease
Brief Title: Impact of Weight Loss Surgery in Adolescents With NAFLD
Acronym: AWLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kathleen E Corey, Director - MGH Fatty Liver Clinic, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014P001504; P30DK040561 (NIH)
Record Dates: First submitted 2016-10-30; First posted 2016-11-02 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: NAFLD; Obesity, Adolescent
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI for steatosis assessment (Experimental): Abdominal MRI for assessment of hepatic steatosis
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI to assess hepatic steatosis

SUMMARY:
This study will assess the impact of weight loss surgery (WLS) on non-alcoholic fatty liver disease (NAFLD) in adolescents as well as the interaction between NAFLD and cardiometabolic risk.

DETAILED DESCRIPTION:
While the impact of WLS has been studied in adults, little is known about NAFLD in adolescents undergoing WLS. At present, only a small number of adolescents undergo WLS each year and thus this area has not been well studied. However, as the prevalence of severe obesity continues to rise the investigators anticipate that so will WLS in adolescents.

This study will establish the impact of WLS on NAFLD in adolescents. Currently, it is assumed that adolescents with NAFLD diagnosed at the time of WLS have universal resolution of their disease with appropriate weight loss, and no further evaluation is conducted. Our group has shown that up to 40% of adolescents who undergo WLS have persistently abnormal aminotransferase levels, suggesting that many may have persistent NASH and are at risk of progressive liver disease. The study will elucidate the history of NAFLD following WLS. Such data have not been previously published and will represent a significant contribution to this field.

ELIGIBILITY:
Inclusion Criteria:

* Obese
* Meets institutional requirements for weight loss surgery

Exclusion Criteria:

* Alcohol consumption or other causes of chronic liver disease
* Intolerance to MRI
* Weight >435 lbs

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in hepatitis steatosis after weight loss surgery | 7 months
  Change in hepatitis steatosis after weight loss surgery as measured by MRS

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Corey, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anticipate to share overall results through publication